CLINICAL TRIAL: NCT01137591
Title: Acetaminophen in Combination With N-Acetylcysteine (NAC) vs. Placebo in the Treatment of Fever: A Double-Blind, Randomized Control Study
Brief Title: Acetaminophen in Combination With N-Acetylcysteine (NAC) Versus Placebo in Treating Fever
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit sufficient participants due to lack of funding; PI has left the institution.
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AAAD4090
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Liver Failure; Liver Failure, Acute; Drug Induced Liver Injury; Prevention & Control; Fever
Keywords: Acetaminophen; Acetylcysteine; Antidotes
MeSH Terms: conditions — Liver Failure; Liver Failure, Acute; Chemical and Drug Induced Liver Injury; Fever | interventions — Acetaminophen; Acetylcysteine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- APAP and NAC combination (Experimental): N-acetyl-p-aminophenol and placebo (APAP-NAC) combination pill
  Interventions: Drug: APAP and NAC combination
- APAP and Placebo combination (Placebo Comparator): N-acetyl-p-aminophenol and placebo (APAP-placebo) combination pill
  Interventions: Drug: APAP and Placebo

INTERVENTIONS:
Drug: APAP and NAC combination — APAP 650mg and NAC 600mg combination oral tablet administered once
  Other Names: APAP: n-acetyl-p-aminophenol; acetaminophen; Tylenol; NAC: n-acetylcysteine; Mucomyst
  Arms: APAP and NAC combination
Drug: APAP and Placebo — APAP 650mg and Placebo combination oral tablet administered once
  Other Names: APAP: n-acetyl-p-aminophenol; acetaminophen; Tylenol
  Arms: APAP and Placebo combination

SUMMARY:
The purpose of this study is to compare the efficacy of the an N-acetyl-p-aminophenol (APAP, also known as acetaminophen) and N-acetylcysteine (NAC) combination versus an APAP-placebo combination as an anti-pyretic agent.

DETAILED DESCRIPTION:
N-acetyl-p-aminophenol (APAP), or more commonly known as acetaminophen in the United States, accounts for more overdose and overdose deaths in the United States and United Kingdom than any other pharmaceutical agent. If N-acetylcysteine (NAC) is given within 8 to 10 hours of APAP ingestion, it has been shown to prevent serious liver failure and death in the setting of overdoses. Therefore, it may be beneficial to administer APAP in combination with NAC routinely to reduce rates of liver failure and death. Because NAC's main role is to reduce the accumulation of APAP's toxic metabolites, the concomitant administration of NAC should have no impact on the efficacy of APAP as an antipyretic and analgesic. Thus, we propose a single-center, non-inferiority randomized control study comparing the efficacy of the APAP-NAC combination as compared to APAP-placebo as an anti-pyretic agent.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 to 75 years old
* admitted to an inpatient unit at Columbia-Presbyterian Medical Center
* fever defined as an oral temperature of 38.5°C

Exclusion Criteria:

* if oral temperature cannot be obtained
* abnormal aminotransferase levels
* prior adverse reaction to acetaminophen or N-acetylcysteine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-04

PRIMARY OUTCOMES:
Difference in temperature reduction between participants who are administered combination N-acetyl-p-aminophenol and N-Acetylcysteine (APAP-NAC) versus combination APAP-placebo | 6 hours after study drug administration

SECONDARY OUTCOMES:
Difference in liver function tests after study drug administration between participants who are administered combination N-acetyl-p-aminophenol and N-Acetylcysteine (APAP-NAC) versus combination APAP-placebo | Within 24 hours of study drug administration
  Change in serum total protein (TP), albumin (Alb), total bilirubin (TB), direct bilirubin (DB), amino alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatate (AP) levels before and after the study drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Chang, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

REFERENCES:
- [Background] Bronstein AC, Spyker DA, Cantilena LR Jr, Green J, Rumack BH, Heard SE. 2006 Annual Report of the American Association of Poison Control Centers' National Poison Data System (NPDS). Clin Toxicol (Phila). 2007 Dec;45(8):815-917. doi: 10.1080/15563650701754763. PMID 18163234
- [Background] Smilkstein MJ, Knapp GL, Kulig KW, Rumack BH. Efficacy of oral N-acetylcysteine in the treatment of acetaminophen overdose. Analysis of the national multicenter study (1976 to 1985). N Engl J Med. 1988 Dec 15;319(24):1557-62. doi: 10.1056/NEJM198812153192401. PMID 3059186
- [Background] Vale JA, Proudfoot AT. Paracetamol (acetaminophen) poisoning. Lancet. 1995 Aug 26;346(8974):547-52. doi: 10.1016/s0140-6736(95)91385-8. No abstract available. PMID 7658783
- See also: Acetaminophen overdose information from the NIH — http://www.nlm.nih.gov/medlineplus/ency/article/002598.htm